CLINICAL TRIAL: NCT04530422
Title: Efficacy of Sofosbuvir Plus Ledipasvir in Egyptian Patients With COVID-19 Compared to Standard Treatment
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Almaza Military Fever Hospital (Other)
Responsible Party: Principal Investigator, Mohamed Abdelsalam El-Gohary, Head of Almaza Military Fever Hospital, Almaza Military Fever Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 14
Record Dates: First submitted 2020-08-26; First posted 2020-08-28 (Actual); Last update posted 2020-08-28 (Actual); Status verified 2020-08

CONDITIONS: Covid19
Keywords: SARS-COV-2; Covid-19; Sofosbuvir- Ledipasvir; Hydroxychloroquine
MeSH Terms: conditions — COVID-19 | interventions — Sofosbuvir; ledipasvir; Oseltamivir; Hydroxychloroquine; Azithromycin

STUDY DESIGN:
Intervention Model Description: This randomized controlled clinical trial is a prospective, comparative, single blind, randomized study that was conducted on 250 patients, divided into two equal groups. The group I received Sofosbuvir plus Ledipasvir and Group II received Oseltamivir, hydroxychloroquine "HCQ" plus Azithromycin (the local medical committee of Almaza Fever Hospital guided standard treatment protocol for COVID-19)
Who Masked: Participant
Masking Description: Randomization applied through computer-generated number and concealed using sequentially numbered, sealed opaque envelope to assign the patient to group 1 either group 2
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- • Group I (Sofosbuvir plus Ledipasvir) (Experimental): Patients assigned to this group (125 patients) were received Sofosbuvir plus Ledipasvir, once daily for 15 to 21 days as minimum and maximum duration of therapy, respectively.
  Interventions: Drug: Sofosbuvir plus Ledipasvir
- Group II (Oseltamivir plus HCQ & Azithromycin) (Active Comparator): Patients in this group (125 patients) were received the local medical committee of Almaza Fever Hospital guided standard treatment protocol for COVID-19:
  * Oseltamivir 150 mg q 12 hours for 10 days ;
  * HCQ 400 q 12 hours for one day followed by 200mg q 12 hours for 9 days ; and
  * Azithromycin 500mg once daily for 1 day , followed by 250mg once daily for 6 days.
  * Additional conservative medications were also given. Patients were evaluated as scheduled on day 0, 5 & 11 clinically
  Interventions: Drug: Sofosbuvir plus Ledipasvir

INTERVENTIONS:
Drug: Sofosbuvir plus Ledipasvir — Sofosbuvir plus Ledipasvir, once daily for 15 to 21days
  * Oseltamivir 150 mg q 12 hours for 10 days ;
  * HCQ 400 q 12 hours for one day followed by 200mg q 12 hours for 9 days ; and
  * Azithromycin 500mg once daily for 1 day , followed by 250mg once daily for 6 days.
  Other Names: Oseltamivir plus Hydroxychloroquine & Azithromycin

SUMMARY:
Currently there is no known effective therapy or vaccine for treatment of SARS-CoV-2, highlighting urgency around identifying effective therapies.

This study aiming to evaluate the anti-HCV medications efficacy "Sofosbuvir-Ledipasvir" in treatment of moderate cases with SARS-COV-2 infection, in comparison to the standard treatment (hydroxychloroquine, oseltamivir and azithromycin).

DETAILED DESCRIPTION:
This randomized controlled clinical trial is a prospective, comparative, single blind, randomized study that was conducted on 250 patients, divided into two equal groups. The group I received Sofosbuvir plus Ledipasvir and Group II received Oseltamivir, hydroxychloroquine "HCQ" plus Azithromycin (the local medical committee of Almaza Fever Hospital guided standard treatment protocol for COVID-19).

Randomization (in RCT only)

Once enrolled in the study, patients randomly assigned to one of the following groups:

* Group I (SL group, n=125): patients received Sofosbuvir plus Ledipasvir.
* Group II (OCH group, n=125): patients received Oseltamivir plus HCQ & Azithromycin.

Randomization applied through computer-generated number and concealed using sequentially numbered, sealed opaque envelope.

Group I Patients assigned to this group (125 patients) were received Sofosbuvir plus Ledipasvir (FDA approved Anti-HCV drug since 2014, with Reference ID: 4081324), once daily for 15 to 21days as minimum and maximum duration of therapy, respectively.

Additional conservative medications were given including, third generation cephalosporines (Ceftriaxone 2 gm /24 hours) for 7 days, methylprednisolone 1 mg/kg/day for 7 days; and prophylactic low molecular weight heparin (enoxaparine) 40 mg/24 hours was given throughout hospitalization period.

Patients were evaluated as scheduled on day 0,5,10 & 15 (also, day 21 if extended duration) clinically, laboratory investigations including RT-PCR & C.T chest. RT-PCR with negative result was repeated after 24-48 hrs.

Medications stopped any time if there was any clinical, radiological or laboratory deterioration.

Group II

Patients in this group (125 patients) were received the local medical committee of Almaza Fever Hospital guided standard treatment protocol for COVID-19:

* Oseltamivir 150 mg q 12 hours for 10 days ;
* HCQ 400 q 12 hours for one day followed by 200mg q 12 hours for 9 days ; and
* Azithromycin 500mg once daily for 1 day , followed by 250mg once daily for 6 days.
* Additional conservative medications were also given. Patients were evaluated as scheduled on day 0, 5 & 11 clinically, laboratory Investigations including RT-PCR & C.T chest. RT-PCR with negative result was repeated after 24-48 hrs. Medication were stopped any time, if there was any clinical, radiological or laboratory deterioration.

2.3 Assessment tools

Basic investigations were applied for all patients on day 0 , repeated on days 5 ,10 & 15 or earlier regarding physician order , including :

* CBC, NLR "neutrophil lymphocyte ratio ".
* ESR.
* AST, ALT, creatinine; fasting blood glucose.
* ECG.
* C.T chest , pneumonia was assessed on admission using CT Severity Scoring System (CT-SSS) and CO-RADS ( Percentage per lobe with max of 5 points for each lobe and 25 points for both lungs ; Right Lung" RUL , RML & RLL " ; Left lung " LUL & LLL " ) (11)

Follow up CT chest was repeated on day 5, 10 and day15 or earlier according to physician's request. It was reported as progressive, regressive, stationary or resolved (progressive: crazy paving +↑CTSS ± consolidation; regressive: i.e. absorption (resolved crazy paving pattern +↓CTSS (12); Cured: complete resolution of pneumonic patches).

Other investigations were asked and repeated when needed including:

* LDH.
* TG.
* D. dimmer.
* S.Ferritin.
* Interleukin 6 level.
* Abdominal U.S.

COVID-19 RT-PCR test was done by extraction of the DNA of the virus by using either device (QIA cube or QIA symphony), it takes 70 minutes for every 12 sample on QIA cube or 5 hours for every 96 samples on the QIA symphony. Then the process was applied for the preparation and implementation of the RT-PCR step by using chemicals for detection of the COVID-19, which takes from one and half hour to two hours for 72 samples.

Discharge criteria

* Resolution of symptoms (Normal body temperature for at least 3 days and significantly improved respiratory symptoms).
* Radiological improvement of pneumonic pattern in CT chest.
* Documented virological clearance in 2 samples at least 24 hours apart.
* There was no co-morbidities or complications, which require hospitalization.
* SpO2 > 93 % without assisted oxygen inhalation.
* Discharge approved by multi-disciplinary medical team.

ELIGIBILITY:
Inclusion Criteria:

* Pneumonic patients with SARS-COV-2 infection confirmed to be positive by RT-PCR; and demonstrated moderate cases criteria (fever "measured temperature of at least 38 °C", lower respiratory symptoms "cough, shortness of breath" and imaging-confirmed pneumonia").
* Female patients enrolled in the study should have no planned pregnancy for 6 months, after participating in the study, with administration of proper contraceptive measures within 30 days from the first therapeutic dose of the investigational drugs.
* Patients agreed to sign an informed consent to participate in the current study and that they would not participate in other clinical trials within 30 days from the last administration of the study drugs.

Exclusion Criteria:

* Severe COVID-19 patients who met one of the following conditions: (1) Respiratory rate (RR) ≥ 30 times / min; (2) SaO2 / SpO2 ≤ 93% in resting state; (3) arterial partial pressure of oxygen (PaO2) / concentration of oxygen (FiO2) ≤ 300 mmHg
* Critical COVID-19 patients with one of the following conditions: (1) respiratory failure and need mechanical ventilation; (2) shock; (3) other organ failure combined with ICU treatment; severe liver disease (such as child Pugh score ≥ C, AST > 5 times upper limit);
* Patients with contraindications specified for sofosbuvir- ledipasvir; the pregnancy test of female subjects during the screening period was positive, the researchers judged that the patient was not suitable to participate in this clinical study due to devastating co-morbid diseases (e.g. de-compensated liver disease, congested heart failure, chronic kidney disease, malignant or hematological disease under therapy or 3 months ago) and patients received antiviral eradication therapy for hepatitis C or B viruses within the previous 6 months.
* Patients with chloroquine contra-indications: QTc > 500 m/sec, myasthenia gravis, porphyria, retinal pathology, epilepsy, G6PD deficiency, allergy to 4-aminoquinolone, chronic heart, kidney or liver disease, and arrhythmias.
* Any patient demonstrates worsening of symptoms, radiological progression with virologically persistence within at least 5 days of the therapeutic evaluation period of the study after exclusion of cytokine storm was considered as a clinical failure and was shifted to the other management protocol.
* Treatment was terminated at any time by a multidisciplinary team if a serious side effect occurred, which was attributed to the medications used ,e.g. cardiac arrhythmia, deteriorated liver or kidney function or unfortunately patient died .

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Actual)
Dates: Start 2020-04-15 (Actual); Primary Completion 2020-07-08 (Actual); Study Completion 2020-07-23 (Actual)

PRIMARY OUTCOMES:
Therapeutic success (cured) | 21 days
  Cured: Documented virological clearance in 2 samples at least 24 hours apart.
28 days in hospital mortality | 28 days
  any incidence of deaths for any participant within 28 days from starting the treatments

SECONDARY OUTCOMES:
Percentage of clinical failure of treatments | 21 Days
  participants who failed to achieve documented virological clearance in 2 samples at least 24 hours apart.
Length of hospital stay | Through study completion, an average of 14 weeks
  days of length of hospital staying in isolation till documented virological clearance in 2 samples at least 24 hours apart.
Incidence of side effects | 21 days
  Incidence of any side effects known to be related to the medication administrated either in group 1 or 2

CONTACTS AND LOCATIONS:
Locations (1):
- Almaza Military Fever Hospital, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No